CLINICAL TRIAL: NCT04477616
Title: Injection Regimen Trial of Pegylated Recombinant Human Granulocyte Colony Stimulating Factor (PEG-rhG-CSF) in Preventing Bone Marrow Suppression and/or Febrile Neutropenia (FN) During Breast Cancer Chemotherapy
Brief Title: Injection Regimen Trial of PEG-rhG-CSF During Breast Cancer Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Jue Wang, Prof., The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NBC Che001
Record Dates: First submitted 2020-07-16; First posted 2020-07-20 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Breast Cancer
Keywords: PEG-rhG-CSF; Bone marrow suppression; Febrile neutropenia; Breast cancer; Chemotherapy
MeSH Terms: conditions — Breast Neoplasms; Febrile Neutropenia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: Experimental/PEG-rhG-CSF (Experimental): patients received a single dose of 6mg of PEG-rhG-CSF(pegfilgrastim), as a single subcutaneous injection on day 7 (chemotherapy day was recorded as day 1). If WBC >= 15 x 10^9/L in the first chemotherapy cycle, then 3mg PEG-rhG-CSF will be used in the second chemotherapy cycle.
  Interventions: Drug: Day 7 regimen
- Comparator: Comparator/PEG-rhG-CSF (Active Comparator): patients received a single dose of 6mg of PEG-rhG-CSF(pegfilgrastim), as a single subcutaneous injection on day 3 (chemotherapy day was recorded as day 1). If WBC >= 15 x 10^9/L in the first chemotherapy cycle, then 3mg PEG-rhG-CSF will be used in the second chemotherapy cycle.
  Interventions: Drug: Day 3 regimen

INTERVENTIONS:
Drug: Day 7 regimen — patients received a single dose of 6mg of PEG-rhG-CSF(pegfilgrastim), as a single subcutaneous injection on day 7 after chemotherapy. If FN occurs in the experimental group and the control group, reduce the dose of chemotherapy in the next course of treatment, timely change the chemotherapy regimen, and closely monitor to ensure patient safety. Record the results of routine blood follow-up and temperature curves of patients at different time periods. If WBC >= 15 x 10^9/L in the first chemotherapy cycle, then 3mg PEG-rhG-CSF will be used in the second chemotherapy cycle.
  Arms: Experimental: Experimental/PEG-rhG-CSF
Drug: Day 3 regimen — patients received a single dose of 6mg of PEG-rhG-CSF(pegfilgrastim), as a single subcutaneous injection on day 3 after chemotherapy. If FN occurs in the experimental group and the control group, reduce the dose of chemotherapy in the next course of treatment, timely change the chemotherapy regimen, and closely monitor to ensure patient safety. Record the results of routine blood follow-up and temperature curves of patients at different time periods. If WBC >= 15 x 10^9/L in the first chemotherapy cycle, then 3mg PEG-rhG-CSF will be used in the second chemotherapy cycle.
  Arms: Comparator: Comparator/PEG-rhG-CSF

SUMMARY:
The purpose of this study is to try to find a better injection regimen (including time and dose) of PEG-rhG-CSF, which is supposed to better prevent bone marrow suppression and/or FN in breast cancer patients who receive chemotherapy.

ELIGIBILITY:
Eligibility Criteria:

1. Female breast cancer aged 18-70 years old, the expected survival period is greater than 12 months.
2. No previous radiotherapy and chemotherapy.
3. No history of serious systemic disease.
4. KPS≥70.
5. White blood cell count> 3.5 × 10 ^ 9 / L, neutrophil count> 1.8 × 10 ^ 9 / L, platelet count> 100 × 10 ^ 9 / L, hemoglobin> 9 g / dl.
6. ALT (alanine transaminase) and AST (aspartate transaminase) <1.5 times the upper limit of normal value, alkaline phosphatase <2.5 times the upper limit of normal value, and total bilirubin <1.5 times the upper limit of normal value.
7. Serum muscle plasma <1.5 times the upper limit of normal value.
8. No abnormal blood coagulation.
9. Women of childbearing age had a negative serum or urine pregnancy test before the start of treatment and agreed to contraception during treatment.
10. Cardiac function: two-dimensional echocardiography examination LVEF (left ventricular ejection fraction) ≥ 55%.
11. Sign informed consent.

Exclusion Criteria:

1. Received systemic or local treatment for tumors, including chemotherapy, radiotherapy, and endocrine therapy.
2. A history of malignant tumors within 5 years (except curable skin basal cell carcinoma and cervical carcinoma in situ).
3. The patient has been enrolled in other clinical trials or used other study drugs 30 days before enrollment in this study.
4. Accompanied by uncontrolled lung disease, severe infection, active gastrointestinal ulcer need treatment, coagulopathy, severe uncontrolled diabetes, connective tissue disease or bone marrow function suppression, and other diseases, can not tolerate chemotherapy-related treatments.
5. Two-dimensional echocardiography detection LVEF <55%.
6. Severe cardiovascular and cerebrovascular diseases within the first 6 months of randomization (eg unstable angina, chronic heart failure, uncontrollable hypertension> 150/90 mmHg, myocardial infarction, or cerebrovascular accident).
7. NCI peripheral neurotoxicity grade ≥2.
8. Those taking glucocorticoids.
9. Known hypersensitivity to anthracyclines, cyclophosphamide, taxanes, trastuzumab, or pertuzumab.
10. Refuse contraception during treatment and within 8 weeks after completion of treatment for women of childbearing age.
11. Pregnant and lactating women.
12. After joining the test, a pregnancy test (+) before using the drug.
13. There are mental illness, cognitive impairment, unable to understand the test plan and side effects, unable to complete the test plan, and follow-up workers (systematic evaluation is required before the trial is enrolled).
14. No personal freedom and independent civil capacity.
15. The investigator determined that the patient could not obtain long-term follow-up data (due to unavailability or serious concomitant diseases).

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2021-07-13 (Actual); Primary Completion 2022-10-06 (Actual); Study Completion 2022-11-06 (Actual)

PRIMARY OUTCOMES:
the rates of grade III/IV neutropenia during the first and second chemotherapy cycle | up to 9 weeks
  grade III or IV neutropenia (ANC < 1x 10^9/L or 0.5 x 10^9/L)
the rates of FN during the first and second chemotherapy cycle | up to 9 weeks
  the occurrent rate of FN（FN：Body temperature ≥38.3°C or ≥38.0°C continued for 1 h, with neutrophil count <500/mcl or neutrophil count <1000/mcl, but expected to drop to <500/ mcl after 48 hours .）

SECONDARY OUTCOMES:
Proportion of patients with down-regulated dosage of PEG-rhG-CSF from 6mg to 3mg | up to 9 weeks
  If WBC >= 10 x 10^9/L in the first chemotherapy cycle, then 3mg PEG-rhG-CSF will be used in the second chemotherapy cycle
Adverse reactions after injection of PEG-rhG-CSF during first and second chemotherapy cycle | up to 9 weeks
  Adverse reactions

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoming Zha, MD, Study Director — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- the First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Xu Y, Huang L, Wang J, He J, Wang Y, Zhang W, Chen R, Huang X, Liu J, Wan X, Shi W, Xu L, Zha X. Exploring optimal administration timing of pegylated recombinant human granulocyte colony-stimulating factor for chemotherapy-induced neutropenia in early breast cancer treated with pharmorubicin and endoxan: a prospective randomized controlled clinical trial. BMC Cancer. 2024 Nov 12;24(1):1387. doi: 10.1186/s12885-024-13156-y. PMID 39533204